CLINICAL TRIAL: NCT01710930
Title: Interest of TARC Serum Marker for Follow-up of Patients With Allergic Broncho-Pulmonary Aspergillosis (ABPA), Excluding Cystic Fibrosis
Brief Title: Protocol TARC-ABPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC11_0158
Record Dates: First submitted 2012-10-15; First posted 2012-10-19 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2017-11

CONDITIONS: Allergic Broncho-Pulmonary Aspergillosis
Keywords: Allergic Broncho-Pulmonary Aspergillosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study of predictive factors (Experimental)
  Interventions: Other: Study of predictive factors

INTERVENTIONS:
Other: Study of predictive factors — Phase 1 : Inclusion of patients (V0) :
  In the case of a participation agreement, data on age, profession, previous history, history of the disease and current treatments will be collected. Different tests will be performed at this visit.
  Phase 2 : Determination of the baseline (V1) : Patients will be reviewed one month after V0 (V1). In the absence of exacerbation between V0 and V1, the examinations performed in routine practice will be used to determine the basic state of biological parameters of interest. During this visit, different tests will be performed.
  Phase 3 : Quarterly monitoring of patients (V2-V9) : Patients will be followed every three months for 2 years (V2-V9).

SUMMARY:
The main objective of this study is to determine if a doubling of serum TARC (compared to baseline) is associated with the occurrence of exacerbations of ABPA.

The secondary objectives of the study are :

1. To investigate if induced sputum eosinophils count (compared to baseline) is associated with the occurrence of exacerbations.
2. To examine if the exhaled NO (compared to a baseline) is associated with the occurrence of exacerbations.
3. To investigate if activation of circulating T cells (compared to a baseline) is associated with the occurrence of exacerbations.
4. To examine if the rate of specific Asp f IgG measured by ELISA (compared to a baseline) is associated with the occurrence of exacerbations.
5. To determine if the variation of one of the markers above, TARC or Asp f specific IgE measured at baseline, may be associated with the radiological stage of the disease (ABPA-S, ABPA-CB, ABPA-ORF).
6. To investigate if there is a link between fungal exposure at home (visually assessed by the contamination level and the proportion of positive samples for Asp. f) and the frequency of exacerbations.
7. To establish if some of the clinical, functional or biological data studied are associated with the frequency of exacerbations.

ELIGIBILITY:
Pre-inclusion criteria :

* Major patients, of indifferent sex,
* Patients insured,
* Patients accepting to give, after information, their signed informed consent form,
* Patients affected by ABPA,
* Patients in remission without treatment, or stable under current treatment for at least 3 months.

Inclusion criteria :

This inclusion will be definitive in V1, if :

* The pre-inclusion criteria are respected,
* The patient has not presented any exacerbation since V0 thereby define a basic state.

If patient could not be included, it will be possible to re-screen him for the study, provided he meets the pre-inclusion and inclusion criteria. In this case, a new V0 will be scheduled at least 3 months after the first V0.

Exclusion criteria :

* Minor patients,
* Adults under guardianship,
* Pregnant or lactating women,
* Patients unable to follow the protocol or to give consent,
* Patients with an infection of the lower respiratory tract in the 4 weeks preceding V0 or between V0 and V1,
* Patients who were hospitalized for respiratory problems in the 4 weeks preceding V0 or between V0 and V1,
* Patients with chronic inflammatory diseases unrelated to ABPA which could influence the results,
* Patients with cancer,
* Patients followed for cystic fibrosis defined by a positive sweat test,
* Patients with known compliance problems identified prior to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-07; Primary Completion 2017-09-21 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
The rate of serum TARC
  The rate of serum TARC will be measured by ELISA and expressed in pg / ml.Doubling of TARC rate compared between baseline (V1) and exacerbations is the primary endpoint (qualitative binary).

SECONDARY OUTCOMES:
Induced sputum eosinophils count
  Increase in induced sputum eosinophils count assessed by cytology between baseline visit (V1) and the visit(s) in exacerbation.
The rate of Exhaled NO(FeNO50)
  Increase in exhaled NO (FeNO50) between baseline visit (V1) and the visit (s) in exacerbation.
The rate of circulating T cells
  Increase in circulating T cells activation, measured by the rate of Th1, Th2, Th17, Treg lymphocytes by flow cytometry before and after specific Asp f. stimulation between baseline visit (V1) and the visit (s) in exacerbation.
The rate of Aspf. specific serum IgG
  Increase of Aspf. specific serum IgG, measured by ELISA between baseline visit (V1) and the visit (s) in exacerbation
Correlation between markers
  Correlation between previous markers, TARC or specific IgE measured at baseline and the stage of the radiological stage of the disease evaluated at V1 (ABPA-S, ABPA-CB, ABPA-ORF).
Fungal exposure at home
  Link of fungal exposure at home with exacerbation frequency and the stage of disease severity.
Clincal parameters
  Link between the clinical parameters (sex, complex aspergillosis, smoking, body mass index, reached ENT associated (chronic rhinitis, sinonasal-polyposis)) and the frequency of exacerbations.
Biological parameters
  Link between the biological parameters measured at stable state (V1) (total IgE, Asp fspecific IgE, Aspergillus precipitins) and the frequency of exacerbations.
Function parameters
  Link between the function parameters measured at baseline state (FEV1 (in%), FVC (in%), compared RV / TLC, FeNO50) and the frequency of exacerbations.

CONTACTS AND LOCATIONS:
Overall Officials: Anaïs PIPET, Doctor, Principal Investigator — Nantes University Hospital; Hakima OUKSEL, Doctor, Study Chair — University Hospital, Angers; François GOUPIL, Doctor, Study Chair — CH du Mans
Locations (2):
- France (2):
  - CHU Le Mans, Le Mans
  - Nantes University Hospital, Nantes